CLINICAL TRIAL: NCT07156110
Title: The Effect of Prosthetic Modality on Bone Level Changes During One-Year Follow-Up
Brief Title: Prosthetic Modality and MBL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Collaborators: Alessio Triestino (Unknown)
Responsible Party: Principal Investigator, Luigi Canullo, professor, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L1
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Bone Loss
Keywords: Marginal bone level changes; prosthetic modalities; soft tissue adaptation
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): Placing Lance+ (Internal Hex connection) implant with a healing abutment. Three months later, after an impression, a screw-retained restoration will be seated using a Ti-Base abutment.
  Interventions: Procedure: Traditional prosthetic procedure
- Arm 2 (Experimental): Placing Lance Conical implant with a healing abutment. Three months later, after an impression, a screw-retained restoration will be seated using a Ti-Base abutment.
  Interventions: Procedure: Traditional prosthetic procedure
- Arm 3 (Experimental): Placing Lance Conical implant together with Connect Abutment (tightened to 30 Ncm) with a Connect healing cap ("one time one abutment"). Screw retained restoration after 3 months.
  Interventions: Procedure: one abutment-one time

INTERVENTIONS:
Procedure: Traditional prosthetic procedure — Three months later, after an impression, haling abutment will be removed and a screw-retained restoration will be seated using a Ti-Base abutment.
  Arms: Arm 1; Arm 2
Procedure: one abutment-one time — Three months later, after an impression, a screw-retained restoration will be seated directly on the connect healing
  Arms: Arm 3

SUMMARY:
The present study will test the effect of different prosthetic modalities on conical and internal hex connection implants, assessing the radiographic MBL changes after one year.

Consecutive patients fulfilling inclusion/exclusion criteria will enter the study. Once the implant is inserted, patients will be divided into three groups according to the time if their inclusion in the study.

Study groups (20 patients per group):

1. Group 1: Placing Lance Conical implant with a healing abutment. Three months later, after an impression, a screw-retained restoration will be seated using a Ti-Base abutment.
2. Group 2: Placing Lance+ (Internal Hex connection) implant with a healing abutment. Three months later, after an impression, a screw-retained restoration will be seated using a Ti-Base abutment.
3. Group 3: Placing Lance Conical implant together with Connect Abutment (tightened to 30 Ncm) with a Connect healing cap ("one time one abutment"). Screw retained restoration after 3 months.

Consecutive inclusion of patients - 1st- group 1, 2nd - group 2, 3rd - group 3 and vice versa.

Primary outcome variable: bone level changes 12 months post-loading

DETAILED DESCRIPTION:
Actually, the histologic composition of the soft tissue around the prosthetic district was Indirectly clarified firstly in animal studies focused on biologic width re- establishment, now renamed supracrestal tissue attachment, which described the epithelial and connective components and the key role in the implant longitudinal maintenance they have (1). In fact, it was shown that the soft tissue morphogenesis in humans may occur in 8-12 weeks (2) This histologic structure is represented by a dense connective tissue with few fibroblasts and edondotelial cells isolated by a junctional epithelium indirectly connected to the abutment in the most coronal portion by a thin layer of proteoglycans and psudopodia (3).

Traditionally the Interaction between living cells and a biocompatible foreign material is mediated by some biological factors and could be associated with a mathematical equation Apparently, this is based on few variables generically represented by soft tissue patterns and biomaterial features (4). In fact, according to the basic science, the host tissue (intended both histologically and epigenetically), the biocompatible foreign material and the antagonist.

The tissue variable should be intended not only as its clinical appearance (thin vs thick), but overall as its INDIVIDUAL regenerative and inflammatory capability (which of course involves also the histologic aspect) (5) Changing our prospecting and focusing on the prosthetic variable, this should be intended not only as it is in its macro/micro and nano structure, but also as it is used in the prosthetic work flow In fact, the proximity of the prosthetic components to the connective tissues (mostly evident in case platform switching configuration) could allow the clinician during the healing period to actively influence soft tissue morphogenesis In fact, 2 weeks after reopening, traditional prosthetic work flow provides for healing abutment disconnection and impression taking (just at the peak of the first phases of wound healing) and two weeks there after new disconnections are required for try ins and definitive prosthetic delivery, just when the maturation healing phase peak occurs(6-7).

These continuous dis-reconnections may lead to soft tissue healing disruption with a long junctional epithelium till the IAJ.

Not to mention the fact that continuous disconnections create a link for the contamination of the connection and the exposure of soft tissues to abutment not always contaminated The only approach able to prevent this "physiological reaction" and allow a complete healing is to adopt a protocol aimed, after an intraoperative impression, to definitively screw the final abutment at the time of second surgery and allow soft tissue to heal undisturbed (so called "one-abutment/one-time) (8) Another factor affecting soft tissue/abutment interaction is the abutment macro design A recent systematic review our group recently produced, suggested that narrower abutments fail to show any difference in terms of soft tissue health (and this is reasonable) and esthetics (9).

On the other hand, the metanalysis highlighted significant differences in terms of MBL in favor of narrower abutments just because this configuration allows for more room for soft tissues supracrestal attachment, probably changing their fiber arrangement from parallel to the long axis to ring-shaped circular with a stronger connective seal Another factor related to the "abutment variable" that dramatically may affect soft tissue/abutment interaction, and therefore interacting with the underlaid bone, is its micro design.

In fact, the importance of the material should be shifted from the bulk to the external surface and its biochemophysical and topographic properties, including cleanliness.

In fact, decontamination of the abutment surface is a prerequisite for cell. Aim The present study will test the effect of different prosthetic modalities on conical and internal hex connection implants, assessing the radiographic MBL changes after one year.

Materials and Methods Study design The study was designed as a prospective, controlled clinical trial with a parallel design. Approval from the Ethics Committee will be obtained before the study commences. Selected patients were informed about the purpose of the study, and if they agreed to participate, they were recruited to participate in the clinical trial once they had signed the informed consent form.

Subject population Subjects in need of an implant-supported restoration will be screened for the following study criteria Consecutive patients fulfilling inclusion/exclusion criteria will enter the study. Once the implant is inserted, patients will be divided into three groups according to the time if their inclusion in the study.

Study groups (20 patients per group):

1. Group 1: Placing Lance Conical implant with a healing abutment. Three months later, after an impression, a screw-retained restoration will be seated using a Ti-Base abutment.
2. Group 2: Placing Lance+ (Internal Hex connection) implant with a healing abutment. Three months later, after an impression, a screw-retained restoration will be seated using a Ti-Base abutment.
3. Group 3: Placing Lance Conical implant together with Connect Abutment (tightened to 30 Ncm) with a Connect healing cap ("one time one abutment"). Screw retained restoration after 3 months.

Consecutive inclusion of patients - 1st- group 1, 2nd - group 2, 3rd - group 3 and vice versa.

Information to collect:

Inclusion day: Demographic data, medical condition Day of surgery: implant site, insertion torque, parallel X-ray. Suture removal - adverse effects. 3 months (impression) - parallel X-ray. Adverse effects. Loading day - parallel X-ray. Adverse effects. 6 months post-loading - parallel X-ray. Adverse effects. 12 months post-loading - parallel X-ray. Adverse effects, pocket depth, BOP.

Clinical photos and videos will be appreciated for future presentations.

Primary outcome variable: bone level changes 12 months post-loading Surgical and prosthetic protocol According to the manufacturer's instructions, using the Lance surgical kit, with tools for Conical connection and internal hex implants (fig 1 and 2).

Prosthetic parts will be inserted according to the manufacturer's instructions using the specific tools and a torque-controlled rachet.

ELIGIBILITY:
Inclusion criteria: 1. Male or female ≥18 years old. 2. One or more adjacent missing teeth in the posterior maxilla or mandible (positions 4-7). A natural tooth had to be present at the mesial end; however, free-end situations were allowed. 3. Adequate bone quality )D1-3) and availability for Lance Conical implant (MIS Implants, Israel) placement of diameters 3.75 mm or 4.2 mm, length 10-13 mm, 4. Patients are willing to participate and attend the planned follow-up visits.

Systemic exclusion criteria: 1. Medical conditions requiring prolonged use of steroids and/or medications that can interfere with bone metabolism. 2. History of leukocyte dysfunction and deficiencies. 3. History of neoplastic disease requiring the use of radiation or chemotherapy. 4. History of renal failure. 5. Metabolic disorders such as osteoporosis. 6. History of uncontrolled endocrine disorders. 7. Physical handicaps that would interfere with the ability to perform adequate oral hygiene. 8. Use any investigational drug or device within 30 days immediately before implant surgery. 9. Alcoholism or any drug abuse. 10. History of immunodeficiency syndromes. 11. Smokers of 10 cigarettes per day, cigar equivalents, or tobacco chewers. 12. In the investigator's opinion, conditions or circumstances would prevent completion of study participation or interfere with the analysis of the study results, such as history of non-compliance or unreliability.

Local exclusion criteria

1. Any bone augmentation performed on the implant site with a healing period of less than 3 months.
2. Local inflammation (including untreated periodontitis).
3. Mucosa disease such as erosive lichen planus
4. History of local irradiation therapy.
5. Presence of osseous lesions
6. History of implant failure
7. Postextraction sites with less than 6 weeks of healing
8. Sever bruxism or cjenching habits
9. Persistent intraoral infection.
10. Bone type 4.

Exclusion criteria at surgery

1. Lack of primary stability less than 35 Ncm.
2. Need for augmentation procedures during implant surgery.
3. Inability to place the implant according to the prosthetic requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MBL | one year post surgery
  magical bone level changes will be measured through X-rays

SECONDARY OUTCOMES:
peri-implant soft tissue variables | one year post surgery
  BoP
peri-implant soft tissue variables | one year post surgery
  Pi
peri-implant soft tissue variables | one year post surgery
  PD

CONTACTS AND LOCATIONS:
Overall Officials: luigi Canullo, prof, Principal Investigator — Studi Odontoiatrici Canullo
Locations (1):
- Studi Odontoiatrici Luigi Canullo, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No
anonymized data will be shared if required